CLINICAL TRIAL: NCT02560389
Title: Dopamine Enhancement of Fear Extinction Learning in PTSD (1R21MH108753)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 204583
Record Dates: First submitted 2015-09-22; First posted 2015-09-25 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Stress Disorder, Post Traumatic
Keywords: Posttraumatic Stress Disorder; functional Magnetic Resonance Imaging; Levodopa (L-DOPA); Exposure Therapy; Fear Extinction
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Levodopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo administered in pill form once by mouth
  Interventions: Drug: Placebo
- 100mg L-DOPA (Active Comparator): 100mg levodopa administered in pill form once by mouth
  Interventions: Drug: Levodopa
- 200mg L-DOPA (Active Comparator): 200mg levodopa administered in pill form once by mouth
  Interventions: Drug: Levodopa

INTERVENTIONS:
Drug: Placebo — Sugar pill packaged to resemble levodopa
  Arms: Placebo
Drug: Levodopa — EIther 100mg or 200 mg, depending on arm assignment, administered once by mouth.
  Other Names: L-DOPA; Larodopa
  Arms: 100mg L-DOPA; 200mg L-DOPA

SUMMARY:
The purpose of this study is to investigate a new use for a medication called levodopa (L-DOPA). L-DOPA has been approved for use in Parkinson 's disease, but not for Posttraumatic Stress Disorder (PTSD). L-DOPA is thought to enhance certain cognitive abilities that the investigators believe may be affected among women with PTSD. It is hypothesized that L-DOPA may enhance fear extinction learning to a conditioned fear stimulus. If this is true, L-DOPA may improve outcomes for those undergoing certain types of therapy for PTSD, though that aim is beyond the scope of this project. Additionally, the investigators are testing whether an individual's genetic profile affects how well L-DOPA works to enhance cognitive abilities.

DETAILED DESCRIPTION:
Current state-of-the art treatments for posttraumatic stress disorder (PTSD) are lacking in efficacy. There are two main evidence-based psychological treatments for PTSD. Prolonged Exposure (PE) is a largely-exposure based intervention that has been found efficacious for the reduction of PTSD symptoms; however, PE is associated with post-treatment remission rates of only ~53-60%. Cognitive Processing Therapy (CPT) is also a widely studied and efficacious psychological treatment for PTSD, which focuses both on exposure to the trauma memory as well as cognitive therapy techniques. As with PE, post-treatment remission rates for CPT are only ~53-60%, thus also indicating need for improvement in overall efficacy and consistency of response across individuals.

There is emerging research demonstrating that dopamine is critical to the consolidation and subsequent recall of fear extinction learning. A recent study of healthy adult humans demonstrated that oral administration of 150 mg L-DOPA after fear extinction learning led to decreased fear responding, even when tested in a new context. Further, this study also found that resting-state functional connectivity, measured ~45 minutes after post-extinction learning L-DOPA administration, between the ventral tegmental area (VTA) and mPFC was correlated with magnitude of medial prefrontal cortex (mPFC) recruitment during recall of the fear extinction learning. This latter finding suggests that the mechanism by which L-DOPA boosts consolidation of fear extinction learning is through acutely reorganized dopaminergic resting-state networks. Indeed, other studies have demonstrated an acute effect of L-DOPA administration on resting-state functional connectivity within dopaminergic neural networks. Thus, agents that increase dopamine transmission acutely during the post-extinction learning consolidation window, and thereby acutely altering organization of dopaminergic neural networks, show promise for boosting the consolidation of fear extinction memories and decreasing fear responding.

Genetic variation is a primary contributor to individual differences in baseline dopamine neurotransmission. Individuals with specific alleles in genes coding for high baseline dopamine demonstrate better performance on tasks probing working memory, cognitive control, and social cognition. Genetic variants in baseline dopamine neurotransmission would therefore be expected to modulate performance-enhancing effects of L-DOPA, such that individuals with low endogenous would be expected to have increased performance upon exogenously increasing dopamine neurotransmission; whereas individuals with high endogenous dopamine would be expected to have performance deteriorate from exogenously increasing dopamine neurotransmission. In support of this hypothesis, a recent study found an interaction between L-DOPA administration and endogenous dopamine neurotransmission (as indicated by a polygenic score pooled across catechol-O-methyltransferase (COMT), dopamine transporter protein (DAT), dopamine D1 receptor (DRD1-3)) on motor learning performance, such that individuals with a combination of alleles coding for higher baseline dopamine demonstrated a weaker learning benefit from L-DOPA, whereas individuals with a combination of alleles coding for lower baseline dopamine demonstrated a stronger learning benefit from L-DOPA. These data demonstrate the non-linear relationship between performance and dopamine levels, suggesting that any investigation of potential effects of boosting dopamine neurotransmission as a means of boosting learning needs to account for baseline dopamine neurotransmission.

Overall, the proposed project seeks to demonstrate the engagement of post-extinction dopamine neurotransmission and downstream acute reorganization of dopaminergic resting-state neural networks as a means of increasing consolidation of generic fear extinction learning in adult women with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* 25-50 years of age
* PTSD related to physical or sexual assault
* Medically healthy
* English speaking

Exclusion Criteria:

* Claustrophobia, or the inability to lie still in a confined space
* Major medical disorders (e.g., HIV, cancer)
* Magnetic metallic implants (such as screws, pins, shrapnel remnants, aneurysm clips, artificial heart valves, inner ear (cochlear) implants, artificial joints, and vascular stents)
* Electronic or magnetic implants, such as pacemakers
* Permanent makeup or tattoos with metallic dyes
* Currently pregnant
* A self-reported history of loss of consciousness (greater than 10 minutes)
* Physical disabilities that prohibit task performance (such as blindness or deafness)
* Psychotic disorders (e.g., schizophrenia)
* Any other condition that the investigator believes might put the participant at risk

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2016-03; Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josh Cisler, PhD., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahrenholtz R, Hiser J, Ross MC, Privratsky A, Sartin-Tarm A, James GA, Cisler JM. Unique neurocircuitry activation profiles during fear conditioning and extinction among women with posttraumatic stress disorder. J Psychiatr Res. 2021 Sep;141:257-266. doi: 10.1016/j.jpsychires.2021.07.007. Epub 2021 Jul 6. PMID 34260994

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 103 participants enrolled but only 91 started in the study. 12 participants did not start in the study (6 did not show up, 3 were claustrophobic, 1 was too large to fit in MRI scanner and 2 were tested positive for having used cannabis)
Period: Overall Study
Arm/Group | Placebo | 100mg L-DOPA | 200mg L-DOPA
Started | 34 | 28 | 29
Completed | 33 | 25 | 27
Not Completed | 1 | 3 | 2
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Tested positive for illicit substance | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 100mg L-DOPA | 200mg L-DOPA | Total
Number analyzed (Participants) | 33 | 25 | 27 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (9) | 35.1 (9.7) | 33.9 (8.4) | 34.23 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 25 | 27 | 85
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 8 | 4 | 15
  White | 25 | 15 | 22 | 62
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 2 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 33 | 25 | 27 | 85

OUTCOME MEASURES:

1. Primary Outcome: Galvanic Skin Response
Description: Differential galvanic skin response will be assessed with respect to the conditioned stimulus versus the control stimulus. The investigators will compare, at an aggregate level, the differential galvanic skin response between the placebo, 100 mg, and 200 mg L-DOPA groups.
Time Frame: Within 30 days of the MRI
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Placebo | 100mg L-DOPA | 200mg L-DOPA
Number analyzed (Participants) | 33 | 25 | 27
Unitless | .37 (0.05) | .29 (0.06) | .36 (0.05)

2. Secondary Outcome: Percentage Change in Functional Activation of Amygdala
Description: Amygdala is the part of the brain which controls emotions, survival instincts, and memory. PTSD patients exhibit hyperactivity in the amygdala in response to stimuli.
  Differential functional activation of the amygdala will be assessed with respect to the conditioned stimulus versus the control stimulus. The investigators will compare, at an aggregate level, the differential functional activation between the placebo, 100 mg, and 200 mg L-DOPA groups.
Time Frame: Within 30 days of the MRI
Population: fMRI data was excluded for following number of participants due to artifacts caused by excessive head motion during the scan.
  Placebo n=4 participants, 100mg L-DOPA n=3 participants, 200mg L-DOPA n=3 participants
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Placebo | 100mg L-DOPA | 200mg L-DOPA
Number analyzed (Participants) | 29 | 22 | 24
Percentage change | -0.1 (0.05) | -0.06 (0.04) | -0.05 (0.04)

3. Secondary Outcome: Functional Activation of Anterior Cingulate Cortex
Description: Differential functional activation of the anterior cingulate cortex will be assessed with respect to the conditioned stimulus versus the control stimulus. The investigators will compare, at an aggregate level, the differential functional activation between the placebo, 100 mg, and 200 mg L-DOPA groups.
Time Frame: Within 30 days of the MRI
Population: Data was excluded for following number of participants due to artifacts caused by excessive head motion during the scan.
  Placebo n=4 participants, 100mg L-DOPA n=3 participants, 200mg L-DOPA n=3 participants
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | 100mg L-DOPA | 200mg L-DOPA
Number analyzed (Participants) | 29 | 22 | 24
percentage change | 0.08 (0.07) | 0.09 (0.04) | 0.07 (0.05)

ADVERSE EVENTS:
Time Frame: 2 days
Description: Non-systematic
Arm/Group | Placebo | 100mg L-DOPA | 200mg L-DOPA
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 0/33 | 0/25 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT02560389/Prot_SAP_000.pdf